CLINICAL TRIAL: NCT04972019
Title: Home-based Virtual Reality System for the Treatment of Chemotherapy-related Cognitive Impairments - Feasibility Study
Brief Title: Telerehabilitation Cognitive Impairments Following Chemotherapy Feasibility Study
Acronym: TCIFCF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bright Cloud International Corp (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Telerehab CH Feasibility; R43CA232936 (NIH)
Record Dates: First submitted 2021-04-07; First posted 2021-07-22 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Impairment, Mild
Keywords: chemotherapy; cognitive impairments; breast cancer; executive functions
MeSH Terms: conditions — Cognitive Dysfunction; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility Sham comparison study:
  Participants are randomized equally into the experimental group and a sham control group. Randomization will be based on a randomization table prepared by a contracted bio-statistician.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will not be told which group the participant is part of, so not be biased in evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation experimental group (Experimental): Experimental training will occur in the home. The experimental training will last 8 weeks, each week having up to 4 sessions of therapeutic game play (based on tolerance). Each session will start with vitals being measured and logged. Data will be uploaded on a secure cloud server to which clinicians will have access.
  Interventions: Device: Telerehabilitation Experimental Group
- Telerehabilitation control group (Sham Comparator): Participants will perform web-based game play while wearing sham equipment. Duration of sessions will be fixed and frequency of sessions will equal that of the experimental group training. Over the total training the control group will have an equal duration of training with the experimental group.
  Interventions: Other: Telerehabilitation Sham Control Group

INTERVENTIONS:
Device: Telerehabilitation Experimental Group — Experimental training will occur in the home. The experimental training will last 8 weeks, each week having up to 4 sessions of therapeutic game play (based on tolerance). Each session will start with vitals and subjective pain level being measured and logged.
  They will wear a computer system modified with biosensors, then do motor and cognitive baselines. Subsequently, participants will play an increasing number of games, targeted at cognitive domains of executive function (primary), memory and attention. At the end of every session vitals and subjective pain will be measured and logged.
  Clinical Coordinator will call homes weekly to ascertain general health and issues with participation.
  At the end of week 4 and 8 participants and their caregivers in the experimental group will fill a subjective evaluation questionnaire to gauge perceived benefits and technical difficulties when using the experimental system. Questions will be scored on a 5-point Likert scale.
  Arms: Telerehabilitation experimental group
Other: Telerehabilitation Sham Control Group — Sham control group will train playing web games while wearing a biosensor connected to a laptop provided, showing the web games. However biosensor data will not be used to control game difficulty.
  Sham group controls will start every session with vitals and subjective pain levels being measured and logged. Then participants will play the same frequency and duration of sessions, however those will consist of web games training the same domains (memory, focusing, executive function). Interaction will be through a mouse, and data will be downloaded to a server maintained by the company doing the web games. Data will then be transferred to the research team.
  At the end of every session vitals and subjective pain levels will again be measured and logged.
  Once a week the Clinical Coordinator will call the home to ascertain general health and determine is there were issues with that week participation.
  Arms: Telerehabilitation control group

SUMMARY:
Develop a game-based upper-extremity motor and cognitive rehabilitation system using custom and adaptable virtual reality simulations on a wearable device enhanced with biosensors.

Participants are stage II and stage III breast cancer survivors with lasting cognitive impairments following their first round of chemotherapy. They will be randomized 1:1 into an experimental group and a sham control group. Each group will train in the home for 8 weeks, during which they will perform up to 4 rehabilitation sessions/week (based on tolerance). Each session will start with vitals being measured and logged. Each group will have three clinical evaluations: 1) at baseline; 2) at 8 weeks post-baseline; and 3) at 16 weeks from baseline for follow up.

Experimental group sessions will consist of increasingly more difficult cognitive training tasks in the form of simulated tasks. Biosensors will be sampled while participants interact with these games while wearing the computer system.

Sham control group will have the same number, suration and frequency of sessions, however they will play web games while wearing some the same biosensors.

Caregivers of all subjects will receive a laptop to be used in filling subjective evaluation forms and sending messages to research team. Training will be in the home, so caregivers will need to support the trials by ensuring compliance with the protocol.

All subjects will undergo standardized clinical evaluations at baseline, at 8 weeks and at 16 weeks from baseline. The subjects in the experimental group will have computerized measures taken during each session, and will fill subjective evaluation forms every 4 weeks of active training.

DETAILED DESCRIPTION:
This portion of the study is intended to provide information pertaining to the feasibility of the experimental system for remote integrative (cognitive and motor) therapy of breast cancer survivors (Stage II or III) with lasting cognitive impairments subsequent to their first chemotherapy regimen, and living in the community with a caregiver.

We aim primarily at determining any clinical benefits in improved cognition (primarily in the executive functions domain), but also increased independence in ADLs, and improved mood (reduced depression). Another outcome is the degree of technology acceptance by the targeted population. Training will be done in the home, thus co-dwelling caregivers will also be recruited.

Specific aims are:

1. testing of a wearable device modified with added biosensors, by breast cancer survivors with CRCI.
2. new technology acceptance and ease of use at home by these individuals;
3. clinical benefit to improved cognition (primarily executive functions and cognitive endurance) when experimental therapy is added to daily routine vs. daily routine plus web-based cognitive games;
4. a therapist console module and enhanced automatic session report that will allow remote monitoring of patient exercising and offline data processing and review.

Participants will be randomized equally in an experimental group, or a sham control group. Experimental subjects will receive computer-based therapy, of increasing duration and intensity for up to 4 sessions/week for 8 weeks. The length of sessions will increase from 15 minutes in week 1 to 40 minutes of actual play in week 8. The longer sessions will also train cognitive endurance, or the ability for sustained cognitive effort. All experimental subjects will have their exercise duration and intensity data logged into the database and investigators will monitor them remotely. An Artificial Intelligence (AI) software layer in the system will progress game difficulty based on success in the games as well as on degree of cognitive engagement, as estimated by the biosensors. Higher cognitive difficulty will be indicative of improved cognition, thus progress in mitigating cognitive impairments subsequent to chemotherapy. Additionally, the duration of training will also be logged, as will be the frequency of training. Longer sessions will be indicative of ability to sustain cognitive engagement longer. Additional input will be obtained from caregivers in the form of periodic questionnaires.

Fatigue will be self-reported during weekly follow up calls by a Clinical Coordinator. Participants will train while seated, and (if needed) their arms can be supported on a table. Rest periods may be introduced as needed, to further mitigate fatigue.

At the end of every other week participants and their caregivers in the experimental group will fill a subjective evaluation questionnaire aimed at gauging perceived benefits and possible technical difficulties when using the BrightGo system. Questions will be scored on a 5-point Likert scale.

Control group will perform an equal amount of web-based game play of assigned cognitive-oriented games.

All participants will undergo screening for cognitive impairments (to confirm Mild Cognitive Impairment at baseline). Then they will continue with their daily routine during their 8-week training, and will undergo a second clinical evaluation at the end of these 8 weeks. All participants will then undergo a third (follow up) evaluation at 8 weeks post-end of training.

Caregivers will support the training by helping ensure compliance to protocol, and will complete subjective evaluation forms to rate the perceive benefit of training for the person they care for.

All participants will receive a weekly call from the Clinical Coordinator so to report on any health concerns and system issues.

ELIGIBILITY:
Recruitment will be at Robert Wood Johnson Medical School and at Rutgers NJ Cancer Institute.

INCLUSION CRITERIA FOR CANCER SURVIVORS WITH CRCI SUBSEQUENT TO CHEMOTHERAPY

* Female breast cancer survivor;
* Age 20 to 65 years;
* At least 12 years of formal education;
* Not participating in other studies;
* Generally healthy and active pre-diagnosis (based on self-report);
* Chemotherapy related cognitive impairments with a Montreal Cognitive Assessment (MoCA) Score 10-25 indicating mild to moderate impairment [Chapman 2016];
* Having had invasive (Stages II and III) breast cancer;
* Had completed standard course of chemotherapy with Anthracyclines: doxorubicin (Adriamycin) & epirubicin (Ellence), or Taxanes: docetalex (Taxotere) & paclitaxel (Taxol), or Combination therapies with like carboplatin, cyclophosphamide (Cytoxan), and fluorouracil (5-FU).
* At least one month post completion of first chemotherapy regimen.
* English speakers so as to comprehend game instructions, feedback forms, clinical exam questionnaires, and neuropsychological testing;
* Adult caregivers male or female can be either spouse, child, or a significant other living in the same home and available for the study;
* Absence of lymphedema or other co-morbidity limiting upper extremity function;
* Low propensity for simulation sickness (as measured by Simulation Sickness questionnaire);
* Living in the community in Central Jersey so to facilitate researchers travel to home for system installation and/or repairs,
* Living with a caregiver willing to support trials and be present during sessions;
* Good upper extremity motor function, able to move arms (at least 30 degrees shoulder, 30 degrees elbow and 30 degrees index finger); 20
* Willing to allow home inspections to ascertain internet conditions in the home, to determine best placement for the experimental system, to install and remove system, and to provide repairs if needed.

EXCLUSION CRITERIA FOR PARTICIPANTS WITH CRCI POST CHEMOTHERAPY

* Male;
* Female participants younger than 20 or older than 65;
* High propensity for simulation sickness (as determined by Simulation Sickness Questionnaire screening);
* Those with severe visual neglect or legally blind;
* Those with severe hearing loss or deafness;
* Those with uncontrolled hypertension (>190/100 mmHg);
* Those with severe cognitive impairment (MoCA score<10);
* Current diagnosis of moderate-severe depression (Beck Depression Inventory II score of 17-63);
* a history of psychiatric illness, defined as serious psychiatric illness such as bipolar mood disorder and schizophrenia, or requiring psychiatric hospitalization.
* a history of or current substance abuse;
* a previous head injury resulting in loss of consciousness;
* a prior diagnosis of neurological illness;
* a current or prior diagnosis of brain cancer;
* non-English speakers;
* Those unable to reliable participate in pre-study assessment due to any reason;
* Those with co-morbidities limiting arm and neck motor function (ex. lymphedema, chronic pain, severe arthritis);
* Less than 1 month post first chemotherapy regimen or starting chemotherapy during 16 weeks post screening (as chemotherapy during study participation is a confounding factor);
* Those with Stage IV (metastatic) breast cancer will be excluded;
* Those presenting with multiple cancers, such as breast and arm bone cancer, or breast and brain cancer;
* Those who are unwilling to allow a home inspection to ascertain Internet quality, determine best placement for the experimental or sham systems, for installation and removal of the systems and necessary repairs.

INCLUSION CRITERIA FOR CAREGIVERS OF PARTICIPANTS WITH CRCI POST CHEMOTHERAPY

* Age 18 or older;
* Generally in good overall health; 21
* Able to converse in English;
* Willing and able to participate in the study;
* Lives with the individual with CRCI post chemotherapy, or comes at least 4 days a week or at least present during home sessions;
* Willing to report on standard of care (e. g. any other treatments during the study) on a weekly basis while enrolled;
* Willing to report on experimental system issues and to fill periodic evaluation questionnaires.

EXCLUSION CRITERIA FOR CAREGIVERS OF INDIVIDUALS WITH CRCI POST CHEMOTHERAPY

* Cardiac, orthopedic, neurologic, psychiatric symptoms limiting participation;
* Dementia;
* Aggressive behaviors (observation);
* Domestic disputes or unstable home environment limiting home based training.

Reasons for exclusion based on these impairments relate to the nature of the virtual rehabilitation training, where participants need to be able to perceive the graphics scene on a head-mounted display, be able to hold game controllers in both hands and interact with therapeutic games, hear the simulation sounds, be aware of their surroundings and be able to sustain rapid arm/fingers movement. While the proposed system is considered safe, malignancies in the upper body, cardiac, orthopedic or neurologic issues can pose bodily risks due to intense activity, risks which we want to minimize. Pregnancy is an exclusion since pregnant women are more prone to simulation sickness. The evaluation instruments are in English, thus subjects who do not speak the language will not comprehend the evaluation questions or instructions, which will bias responses.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female will be recruited, as this study targets breast cancer survivors.
Enrollment: 40 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) | Change from Screening at baseline, to 8 weeks and to 16 weeks from baseline
  Measure of change in cognitive impairment for cancer survivors and their caregivers
Change in Test of Pre-morbid Functioning | Change from baseline, to 8 weeks and to 16 weeks from baseline
  Measure cognitive ability [Pearson Education 2017]
Change in NAB Attention Module | Change from baseline, to 8 weeks and to 16 weeks from baseline
  Measure of sustained attention [Hartman 2006]
Change in NAB Functioning Word Module | Change from baseline, to 8 weeks and to 16 weeks from baseline
  Measure of word generation [White and Stern 2003]
Change in Trail Making Test | Change from baseline, to 8 weeks and to 16 weeks from baseline
  A measure of executive functioning [Raitan 1958]
Change in Hopkins Verbal Learning Test Revised | Change from baseline, to 8 weeks and to 16 weeks from baseline
  Verbal/auditory memory test [Brandt 1991];
Change in Brief Visuo-spatial Memory Test, Revised (BVMT-R) | Change from baseline, to 8 weeks and to 16 weeks from baseline
  Visual memory test [Benedict et al., 1996];

SECONDARY OUTCOMES:
Change in Quality of Life Patient/Cancer Survivor Version (QOL-CSV) | Change from baseline, to 8 weeks and to 16 weeks from baseline
  Quality of Life for Cancer Patients [Ferrell, et al 2012]. Form includes 41 items representing the four domains of quality of life incorporating physical, psychological, social, and spiritual well being.
  Each question is scored on a 0 to 10 scale.
Caregiver Quality of Life-Cancer (CQOL-C) | Change from baseline, to 8 weeks and to 16 weeks from baseline
  Questionnaire for caregiver oncology quality of life [Weitzner et al 1999]
Change in Beck Depression Inventory II | Change from baseline, to 8 weeks and to 16 weeks from baseline
  Measure of depression severity [Beck 1996]
Change in Grasp strength (Jamar dynamometer) | Change from baseline to 8 weeks and to 16 weeks from baseline
  measure of sustained grasping force
Change in Shoulder strength (wrist weights) | Change from baseline, to 8 weeks and to 16 weeks from baseline
  measure of sustained shoulder strength
Change in Range of motion (goniometer) | Change from baseline, to 8 weeks and to 16 weeks from baseline
  measure of upper extremity range of motion
Change in Jebsen test of hand function | Change from baseline, to 8 weeks and to 16 weeks from baseline
  Timed battery of simulated ADLs
Change in Chedokee test (CAHAI-9) | Change from baseline, to 8 weeks and to 16 weeks from baseline
  Timed battery of simulated bimanual ADLs
Change in Game performance | Change in daily performance during 8 weeks experimental therapy
  Objective measure of participant performance in the therapeutic games.
Change in Subjective evaluation questionnaire | change in scores at 4 weeks and at 8 weeks from baseline
  subjective evaluation on a Likert scale of system and perceived benefits by participant and by caregiver
biosensor data | at every session during 8 weeks experimental therapy following baselining
  measure of skin conductance (indicative of sweat) as an indirect indication of cognitive engagement, blinking rate and gaze.
Change in Subjective Pain Rating Scale | Change in subjective pain rating score from baslie to end of 8 weeks experimental therapy and at evaluation sessions
  10-point scale rating pain severity

OTHER OUTCOMES:
Cyber-sickness Susceptibility Questionnaire for participant | Screening at consent
  Form used at screening post-consent to determine a participant's propensity for simulation sickness [Freiwald et al., 2020]. The questionnaire asks participants 26 questions The first 13 questions ascertain the general heath and fitness of the subject, and have Yes/No answers The remaining 13 questions are score on a on a 5 point Likert scale, with five point Likert scales, referring to the frequency of each complaint's occurrence. These scales range from 0 to 4 with the labels "very rarely", "rarely", "occasionally", "frequently" and "very often".
Change in Heart rate | Change in heart rate from baseline to end of 8 week trainig measured every session.
  Heart rate (Pulse) measured with a medical meter at start and end of each training session
Change in Blood pressure (systolic and diastolic) | Change in heart rate from baseline to end of 8 week trainig measured every session.
  Blood pressure (systolic and diastolic) measured with a medical meter at start and end of each training session

CONTACTS AND LOCATIONS:
Overall Officials: Grigore C Burdea, PhD, Principal Investigator — Bright Cloud Int'l Corp
Locations (2):
- United States (2):
  - Rutgers University Rober Wood Johnson Medical School, New Brunswick, New Jersey
  - Bright Cloud Int'l Corp, North Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymized and made available through scientific publications.
Supporting Information: ICF
Time Frame: After completion of study